CLINICAL TRIAL: NCT03230994
Title: A Study of Cooperative Network of Diagnosis and Treatment of Uterine Adenomyosis.
Brief Title: Cooperative Adenomyosis Network
Acronym: CAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Aijun Sun, Professor, Peking Union Medical College Hospital
Other Study IDs: CAN201706
Record Dates: First submitted 2017-06-30; First posted 2017-07-27 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Dysmenorrhea; Metrorrhagia; Infertility, Female; Pathology; Ultrasonography; Radiography
Keywords: adenomyosis; diagnosis; treatment; epidemiology; Complications
MeSH Terms: conditions — Dysmenorrhea; Metrorrhagia; Infertility, Female; Adenomyosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Different Treatment Groups: Women would receive different pharmacotherapy from the standard approach，such as levonorgestrel-releasing intrauterine system(LNG-IUS)，Gonadotrophin releasing hormone agonist(GnRH-a),surgery,etc.

SUMMARY:
To set up a Cooperative Network by enrolling 5000 patients with Adenomyosis(AM) from multiple centers.Based on the Network platform and Database,the investigators try to explore the diagnostic strategies for AM and carry out epidemiological survey on the semeiology of AM.In addiction，the investigators expect to conduct research on the effect and the follow-up fertility outcomes of different medical or surgical treatment, the etiology of AM and endometriosis,the perspective investigation of the malignant transformation of AM ;the high-risk factors of AM,and finally propel the formation of Expert Consensus and Clinical Guidelines about AM which suitable to chinese conditions.

DETAILED DESCRIPTION:
5000 women diagnosed of Adenomyosis(AM) with pathology, transvaginal ultrasonography or magnetic resonance image（MRI）will be enrolled from nationwide multicenters. The investigators would build up Network platform, and database with the registered data within 6 months. 30-month follow-up with an interval of at least once every 6 months will be done for every patient ，and update the database timely.

Based on the Network platform and Database,we try to explore the diagnostic strategies for AM and carry out epidemiological survey on the semeiology of AM.In addiction，the investigators expect to conduct research on the effect and the follow-up fertility outcomes of different medical or surgical treatment,the etiology of AM and endometriosis,the perspective investigation of the malignant transformation of AM ;the high-risk factors of AM,and finally propel the formation of Expert Consensus and Clinical Guidelines about AM which suitable to chinese conditions.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed of adenomyosis by pathology, transvaginal ultrasound or MRI.

Exclusion Criteria:

* Refusal to join the study

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: 5000 women diagnosed of adenomyosis by pathology or magnetic resonance image（MRI）by experienced specialist physicians will be enrolled from nationwide multicenter.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effect and Diagnostics | 2day
  Symptom Assessment

SECONDARY OUTCOMES:
Pathology | 1day
  Diagnostic assessment
selection of therapeutic scheme | 1day
  pharmacotherapy or surgery
vision algetic standard（VAS） | 2day
  Semeiology and evaluative criteria
B type ultrasound | 1day
  Diagnostic assessment
Magnetic Resonance Imaging | 1day
  Diagnostic assessment
pictorial blood loss assessment chart（PBAC） | 2day
  Semeiology and evaluative criteria

CONTACTS AND LOCATIONS:
Overall Officials: Aijun AJ SUN, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Lei Li, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: Yes
Network platform, and the website will be attached later.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Within twelve months after the trial complete
Access Criteria: Data access requests will be reviewed by an external independent review panel.Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Struble J, Reid S, Bedaiwy MA. Adenomyosis: A Clinical Review of a Challenging Gynecologic Condition. J Minim Invasive Gynecol. 2016 Feb 1;23(2):164-85. doi: 10.1016/j.jmig.2015.09.018. Epub 2015 Sep 30. PMID 26427702
- [Background] Alabiso G, Alio L, Arena S, Barbasetti di Prun A, Bergamini V, Berlanda N, Busacca M, Candiani M, Centini G, Di Cello A, Exacoustos C, Fedele L, Fuggetta E, Gabbi L, Geraci E, Imperiale L, Lavarini E, Incandela D, Lazzeri L, Luisi S, Maiorana A, Maneschi F, Mannini L, Mattei A, Muzii L, Pagliardini L, Perandini A, Perelli F, Pinzauti S, Porpora MG, Remorgida V, Leone Roberti Maggiore U, Seracchioli R, Solima E, Somigliana E, Tosti C, Venturella R, Vercellini P, Vigano P, Vignali M, Zannoni L, Zullo F, Zupi E; Endometriosis Treatment Italian Club. Adenomyosis: What the Patient Needs. J Minim Invasive Gynecol. 2016 May-Jun;23(4):476-88. doi: 10.1016/j.jmig.2015.12.017. Epub 2016 Jan 6. PMID 26772777
- [Result] Vercellini P, Consonni D, Barbara G, Buggio L, Frattaruolo MP, Somigliana E. Adenomyosis and reproductive performance after surgery for rectovaginal and colorectal endometriosis: a systematic review and meta-analysis. Reprod Biomed Online. 2014 Jun;28(6):704-13. doi: 10.1016/j.rbmo.2014.02.006. Epub 2014 Mar 4. PMID 24745831
- [Result] Pontis A, D'Alterio MN, Pirarba S, de Angelis C, Tinelli R, Angioni S. Adenomyosis: a systematic review of medical treatment. Gynecol Endocrinol. 2016 Sep;32(9):696-700. doi: 10.1080/09513590.2016.1197200. Epub 2016 Jul 5. PMID 27379972
- [Result] Li L, Leng JH, Shi JH, Zhang JJ, Jia SZ, Li XY, Dai Y, Zhang JR, Li T, Xu XX, Liu ZZ, You SS, Chang XY, Lang JH. [A prospective study on the effects of levonorgestrel-releasing intrauterine system for adenomyosis with menorrhagia]. Zhonghua Fu Chan Ke Za Zhi. 2016 Jun 25;51(6):424-30. doi: 10.3760/cma.j.issn.0529-567X.2016.06.005. Chinese. PMID 27356477
- [Result] Sakhel K, Abuhamad A. Sonography of adenomyosis. J Ultrasound Med. 2012 May;31(5):805-8. doi: 10.7863/jum.2012.31.5.805. No abstract available. PMID 22535729
- [Result] Levy G, Dehaene A, Laurent N, Lernout M, Collinet P, Lucot JP, Lions C, Poncelet E. An update on adenomyosis. Diagn Interv Imaging. 2013 Jan;94(1):3-25. doi: 10.1016/j.diii.2012.10.012. Epub 2012 Dec 12. PMID 23246186
- [Derived] Chen X, Lang J, Li L. Adenomyosis Patterns on Transvaginal Sonography Could Predict the Obstetrical Outcomes of Fertility-Sparing Surgeries: A Retrospective Cohort Study. J Minim Invasive Gynecol. 2025 Jun;32(6):540-549. doi: 10.1016/j.jmig.2025.01.003. Epub 2025 Jan 11. PMID 39805535
- See also: Clinical Challenge — https://www.ncbi.nlm.nih.gov/pubmed/?term=Adenomyosis%3A+A+Clinical+Review+of+a+Challenging+Gynecologic+Condition.
- See also: Treatment Choices — https://www.ncbi.nlm.nih.gov/pubmed/?term=Adenomyosis%3A+What+the+Patient+Needs.+J+Minim+Invasive+Gynecol.
- See also: Fertility Outcome — https://www.ncbi.nlm.nih.gov/pubmed/?term=Adenomyosis+and+reproductive+performance+after+surgery+for+rectovaginal+and+colorectal+endometriosis%3A+a+systematic+review+and+meta-analysis.
- See also: Medical Treatment — https://www.ncbi.nlm.nih.gov/pubmed/27379972
- See also: ING-IUS — https://www.ncbi.nlm.nih.gov/pubmed/27356477
- See also: Transvaginal Sonography — https://www.ncbi.nlm.nih.gov/pubmed/?term=Sonography+of+adenomyosis.+J+Ultrasound
- See also: MRI — https://www.ncbi.nlm.nih.gov/pubmed/?term=An+update+on+adenomyosis.+Diagn+Interv+Imaging

DOCUMENTS (2):
  • Informed Consent Form (2017-06-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT03230994/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-06-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT03230994/Prot_SAP_001.pdf